CLINICAL TRIAL: NCT04106869
Title: Does Intra-operative Low End Tidal CO2 Aggravate Perioperative Neurocognitive Disorders?
Brief Title: The Influence of Ventilation on Perioperative Neurocognitive Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution and the study was not continued
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Principal Investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Venti-delirium
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be blinded to the group, as well as the outcomes assessor and the investigator.
  The anesthesiologist responsible for the patient's anesthesia will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperventilation (Active Comparator): Ventilatory settings will be the following:
  6-8 ml/kg and Respiratory rate adjusted to the required ETC02 (<35 mmHg) PEEP in order to ensure a driving pressure (P plateau- PEEP) below 15 mmHg.
  Interventions: Other: Hyperventilation
- Hypoventilation (Placebo Comparator): Ventilatory settings will be the following:
  6-8 ml/kg and Respiratory rate adjusted to the required ETC02 ( 40-45 mmHg) PEEP in order to ensure a driving pressure (P plateau- PEEP) below 15 mmHg.
  Interventions: Other: Hypoventilation

INTERVENTIONS:
Other: Hyperventilation — Ventilatory settings will be the following:
  6-8 ml/kg and Respiratory rate adjusted to the required ETC02 (<35 mmHg) PEEP in order to ensure a driving pressure (P plateau- PEEP) below 15 mmHg.
  Arms: Hyperventilation
Other: Hypoventilation — Ventilatory settings will be the following:
  6-8 ml/kg and Respiratory rate adjusted to the required ETC02 (40-45 mmHg) PEEP in order to ensure a driving pressure (P plateau- PEEP) below 15 mmHg.
  Arms: Hypoventilation

SUMMARY:
This prospective study is designed to examine the influence of intra-operative ventilation on perioperative neurocognitive disorders in patients undergoing total hip arthroplasty.

DETAILED DESCRIPTION:
Perioperative neurocognitive disorders (PND's) remain an important complication after surgery. After many years of speculating about the etiology of this complication, currently studies are pointing to an inflammatory cascade being set in motion. Following the combination of surgery/ anesthesia, high molecular group box protein 1 (HMGB1) is released. This damage-associated molecular pattern (DAMP) binds to pattern recognition receptors (PRR) on circulating bone marrow-derived monocytes (BM-DMs). Through an intracellular signaling pathway, the transcription factor NF-kappa B passes into the nucleus, is activated and increases expression and release of pro-inflammatory cytokines. These in turn disrupt the blood brain barrier. Within the brain parenchyma the chemokine monocyte chemoattractant protein 1 (MCP-1) is upregulated and attracts the BM-DMs through binding to its receptor, CCR2. In turn, this activates the resident quiescent microglia. Together, the BM-DMs and activated microglia release HMGB1 and pro-inflammatory cytokines that disrupt long-term potentiation (LTP) thereby blocking synaptic plasticity changes that are required for the cognitive functions of learning and memory.

Optimizing intraoperative ventilation has been the goal of many studies, which have suggested obtaining protective ventilation through the use of low tidal volumes (6-8 ml/kg) and driving pressure below 15 mm Hg.

Very few articles have focused on the influence of intra-operative ventilatory management on PND's.

This prospective study is designed to examine the influence of intra-operative ventilation on perioperative neurocognitive disorders in patients undergoing total hip arthroplasty.

The objectives in our study are to:

Evaluate the influence of intra-operative ventilation on the incidence of incidence and duration of perioperative neurocognitive disorders in a known high-risk group of surgical patients.

Measure peripheral inflammatory markers (IL-6) in the same group of surgical patients.

The evaluation of the presence of peri-operative neurocognitive disorders in patients scheduled for a total hip arthroplasty will be done by using the T-MOCA test. Patients will have to take this test at three time-points (Baseline, 6 weeks post-operatively and 3 months post-operatively.) Patients will be randomized to two groups. One group will be ventilated to obtain intra-operative end-tidal CO2 below 35 mm Hg and the other group will be ventilated to obtain intra-operative end-tidal CO2 of 40-45 mm Hg. Peripheral inflammatory markers will as well be measured in the same group of patients.

Anesthesia management of these patients will comply to our hospital's standard of care practice.

Monitoring of Physiological Parameters During General Anesthesia: Heart rate, oxygen saturation (SpO2), respiratory rate, non-invasive blood pressure, end-tidal CO2 levels, inspired/end-tidal O2 levels, inspired/end-tidal sevoflurane concentrations, and temperature will be continuously monitored and recorded throughout the surgical procedure, to ensure that the measured physiological parameters are within the normal range.

Similarly, the cumulative doses of all sedative and analgesic medications will also be recorded.

Induction and Maintenance of General Anesthesia:

All patients will receive general anesthesia using an endotracheal tube to facilitate ventilatory support.

Induction of anesthesia will be performed using the following:

I.V. Sufentanil 0.1- 0.2 mcg/kg I.V. Lidocaine 1.5 mg/kg I.V. Propofol 2-3 mg/kg I.V. Rocuronium 0.6 -1.2 mg/kg General anesthesia will be maintained using 0.5-2.5% sevoflurane in an O2:air mixture.

Ventilatory settings will be the following:

6-8 ml/kg and Respiratory rate adjusted to the required ETC02 (end-tidal C02) PEEP (positive end-expiratory pressure) in order to ensure a driving pressure (P plateau- PEEP) below 15 mmHg Additional analgesia will be provided with I.V. Acetaminophen 15 mg/kg and I.V. Diclofenac 1 mg/kg, I.V. Tramadol 1-2 mg/kg and, if necessary, additional boluses of I.V. sufentanil 5 mcg.

If muscle relaxation is required by the surgeon, I.V. rocuronium may be administered in 10-20 mg boluses. I.V. Sugammadex 4 mg/kg will be administered if needed to reverse neuromuscular blockade.

Upon emergence from anesthesia:

All patients will be transferred to the post-operative recovery unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ASA (American Society of Anesthesia) score of I- III
* Scheduled for total hip arthroplasty

Exclusion Criteria:

* lack of local language comprehension
* neuropsychiatric disturbance
* history of drug/alcohol abuse
* use of anticholinergic drugs, benzodiazepines, opiates/neuroleptic drugs
* patients with an infectious disease within the last month/immune-suppressant therapy within the last 2 months (e.g., azathioprine or cyclosporine) or chronic medication with potential immune-modulatory effects
* patients who underwent major surgery within the last 3 months
* Patients with cardiovascular, or respiratory diseases (including smoking) resulting in clinically relevant impaired function
* Patients with pre-existing CVA, dementia, and other neurological conditions that would interfere with their ability to participate cognitively
* patients with active malignancy

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
T-MOCA-baseline | 12 hours
  In order to evaluate perioperative neurocognitive disorders, patients will take the T-MOCA test
T-MOCA-6-weeks-postoperatively | 6 weeks
  In order to evaluate perioperative neurocognitive disorders, patients will take the T-MOCA test
T-MOCA-3-months-postoperatively | 3 months
  In order to evaluate perioperative neurocognitive disorders, patients will take the T-MOCA test

SECONDARY OUTCOMES:
Concentration of patient's baseline pre-operative peripheral IL-6 | 12 hours
  Blood samples to measure IL-6 will be drawn prior to the surgery
Concentration of patient's post-operative peripheral IL-6; 6 hours post-operative | 24 hours
  Blood samples to measure IL-6 will be drawn 6 hours after the surgery
Concentration of patient's post-operative peripheral IL-6 ; 24 hours post-operative | 24 hours
  Blood samples to measure IL-6 will be drawn 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Saxena, MD, Principal Investigator — CHU Charleroi
Locations (1):
- CHU-Charleroi Hopital Civil Marie Curie, Charleroi, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No